CLINICAL TRIAL: NCT01548560
Title: Assessing the Safety of Dapivirine Gel and Film Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FAME 02; NCT01662245 (obsolete NCT alias)
Record Dates: First submitted 2012-03-01; First posted 2012-03-08 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections
Keywords: HIV Infections; Anti-HIV agents; HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Dapivirine Vaginal Gel (Experimental): Dosage form: vaginal gel Dosage: 0.5%, 2.5g Frequency: 7 daily doses
  Interventions: Drug: Dapivirine Vaginal Film; Drug: Dapivirine Vaginal Gel
- Placebo Gel (Placebo Comparator): Dosage form: vaginal gel Dosage: N/A Frequency: 7 daily doses
  Interventions: Drug: Dapivirine Vaginal Gel
- Dapvirine Vaginal Film (Experimental): Dosage form: vaginal film Dosage: 1.25mg Frequency: 7 daily doses
  Interventions: Drug: Dapivirine Vaginal Film; Drug: Dapivirine Vaginal Gel
- Vaginal Film (Placebo Comparator): Dosage form: vaginal film Dosage: N/A Frequency: 7 daily doses
  Interventions: Drug: Dapivirine Vaginal Film

INTERVENTIONS:
Drug: Dapivirine Vaginal Film — Dosage form: vaginal film Dosage: 1.25mg Frequency: 7 daily doses
  Arms: Dapivirine Vaginal Gel; Dapvirine Vaginal Film; Vaginal Film
Drug: Dapivirine Vaginal Gel — Dosage form: vaginal gel Dosage: 0.5%, 2.5g Frequency: 7 daily doses
  Arms: Dapivirine Vaginal Gel; Dapvirine Vaginal Film; Placebo Gel

SUMMARY:
This is a study to determine the safety of dapivirine gel and dapvirine film for healthy, HIV-uninfected women aged 18-45 years using the product for 7 daily doses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 45 years (inclusive) at screening
* Able and willing to provide written informed consent to be screened for and to take part in the study.
* Able and willing to provide adequate locator information
* HIV-uninfected based on testing performed by study staff at screening (per algorithm in Appendices I)
* Per participant report, using an effective method of contraception at enrollment; hormonal method (except vaginal ring) used continuously for the past 30 days; intrauterine device (IUD inserted at least 30 days prior to enrollment); female sterilization; abstinent from sexual activity with male partner for the past 30 days; or sexual activity with vasectomized partner; and willingness to use effective method of contraception until the completion of final scheduled study visit if enrolled (approximately 35 days after enrollment)
* In general good health as determined by the site clinician
* For participants older than 21, a pap result in the 12 calendar months prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009) or satisfactory evaluation with no treatment required of non-Grade 0 Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines or per local standard of care, in the 12 calendar months prior to the Enrollment

Note: For participants aged 18-21, a Grade-0 or adequately evaluated abnormal Pap smear is not required as the American Society for Colposcopy and Cervical Pathology recommends initiating screening at age 21.

* Agree to be sexually abstinent from Visit 1 until the completion of Visit 3
* Agree to use study condoms between Visits 3 and 4 (if heterosexually active)
* Agree to abstain from any other intravaginal product or penetration (including sex toys, excluding tampons) until Visit 3
* Willingness to undergo all study-related assessments and follow all study-related procedures
* At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial

Exclusion Criteria:

* Menopause (as defined as amenorrhea for one year or more without an alternative etiology)
* Hysterectomy
* Participant report of any of the following:

  * Known adverse reaction to any of the study products (ever)
  * Known adverse reaction to latex (ever)
  * Non- therapeutic injection drug use in the 12 months prior to Screening
  * Surgical procedure involving the pelvis in the 90 days prior to enrollment (includes dilation and curettage or evacuation, and cryosurgery; does not include cervical biopsy for evaluation of an abnormal pap smear)
  * Participation in a drug, spermicide and/or microbicide study in the 30 days prior to enrollment or anticipated participation in an investigational drug study in the next 8 weeks
  * Pregnancy within 90 days of enrollment
  * Currently lactating
  * Use of a diaphragm, NuvaRing®, or spermicide for contraception
  * Internal vaginal use of any device or product (except tampons) in the 7 days prior to enrollment
* Urogenital infection or suspected infection within 14 days of enrollment including: symptomatic candidiasis, trichomonas vaginalis, and symptomatic bacterial vaginosis; or cervical infection, including N. gonorrhea, C. trachomatis, or mucopurulent cervicitis; syphilis; HSV lesions, or other sores (Note: seropositive HSV without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection; recent exposure to a partner with GC, CT, Trichomonas, syphilis, or NGU
* Antibiotic or antifungal therapy (vaginal or systemic) within 7 days of enrollment
* As determined by the PI, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
* Menses or other vaginal bleeding at the time of the Enrollment visit
* Has any of the following laboratory abnormalities per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0 December 2004:

  * Grade 1 or higher AST or ALT
  * Grade 1 or higher creatinine
  * Grade 2 or higher hemoglobin
  * Grade 1 or higher platelets (Note: otherwise eligible participants with an exclusionary test may be re-tested during the screening process).
* Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of Grade 2 or higher Adverse Events | 5-11 weeks
  The safety/toxicity endpoint is clinical or laboratory evidence of a Grade 2 or higher Adverse Event as defined by the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 and the Female Genital Grading Table for Use in Microbicide Studies which is judged to be related to study product.

SECONDARY OUTCOMES:
Changes in vaginal flora and vaginal pH | 5-11 weeks
Systemic and local absorption levels of dapivirine | 5-11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD MPH, Study Chair — Magee Womens Hospital, UPitt
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States